CLINICAL TRIAL: NCT02782572
Title: Safety and Efficacy of Exercise Training in Patients With Acute Heart Failure: a Pilot Study
Brief Title: Safety of Aerobic Exercise in Acute Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Mayron Faria de Oliveira, PhD, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3646
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure; Acute Heart Failure
Keywords: Exercise; Cardiac Rehabilitation; Non-invasive ventilation
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise; Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise with Non-invasive ventilation (Experimental): Patients with acute haert failure who performed aerobic exercise with non-invasive ventilation. This group also received conventional medical treatment.
  Interventions: Other: Exercise
- Exercise (Sham Comparator): Patients with acute haert failure who performed aerobic exercise with placebo of non-invasive ventilation. This group also received conventional medical treatment.
  Interventions: Other: Exercise
- Control (Other): Patients who receiveid only conventional medical treatment and not performed exercise during protocol.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise in acute heart failure in three different groups (conventional medical treatment; exercise with non-invasive ventilation and exercise with placebo of non-invasive ventilation).
  Other Names: Conventional medical treatment; Non-invasive ventilation

SUMMARY:
This project deals with exercise in acute heart failure in three different groups (conventional medical treatment; exercise with non-invasive ventilation and exercise with placebo of non-invasive ventilation).

DETAILED DESCRIPTION:
All of the subjects performed an individualized clinical evaluation right after hospital admission on day 1 (D1) by the cardiologist and physiotherapis involved in the study. Pulmonary function tests (spirometry), blood sample (brain natriuretic peptide [NT-proBNP] and high sensitive C-reactive protein [hs-CRP]), six-minute walk test (6MWT), and maximal inspiratory pressure (MIP) test were performed.

After the clinical tests were performed, the patients were randomized into three groups, and all received standard medical treatment.

The control group (CTL) received medical treatment and did not perform aerobic exercise training; the ET+NIV group performed aerobic exercise training associated with NIV once a day, for 8 consecutive days; and the ET+Sham group performed aerobic exercise with placebo NIV once a day, for 8 consecutive days. The ET+NIV and ET+Sham groups also received medical treatment.

After eight consecutive days, all of the patients underwent a new clinical evaluation (D10). After D10, all of the patients continued to receive only conventional treatment, and they were followed up for main outcomes (hospital discharge, worsening HF, or death). Worsening HF was considered when a patient needed to be transferred to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of acute HF; previous Doppler echocardiography with left ventricle ejection fraction (LVEF) <30%, and NYHA Class IV.

Exclusion Criteria:

* unstable angina, complex cardiac arrhythmias, pacemaker, cardiac resynchronization therapy or left ventricle assist device, myocardial infarction within the previous 12 months, oxygen saturation by pulse oximetry (SpO2) at rest < 88% without oxygen supplementation, acute pulmonary edema with clinical indications for mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of exercise in acute heart failure | Patients were followed up until hospital discharge. up to 60 days
  After exercise protocol, all of the patients continued to receive only conventional treatment, and they were followed up for main outcomes (hospital discharge, worsening HF, or death). Worsening HF was considered when a patient needed to be transferred to the intensive care unit.

IPD SHARING:
Plan to Share IPD: No